CLINICAL TRIAL: NCT00479089
Title: Phase II Trial of Weekly Docetaxel (Taxotere) Vs. Weekly Docetaxel in Combination With ZD1839 (Iressa®) As Consolidation Therapy For Metastatic Urothelial Cancer Following Maximal Response To Multi-Agent Chemotherapy
Brief Title: Iressa and Taxotere Study in Patients With Metastatic Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted due to drug sponsor decision to not continue.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0767; NCI-2010-00595 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-09

CONDITIONS: Bladder Cancer
Keywords: Transitional Cell Carcinoma; Urothelium; Urothelial Cancer; Bladder Cancer; Docetaxel; Taxotere; ZD1839; Gefitinib; Iressa; Consolidation Therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Docetaxel; Gefitinib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weekly Docetaxel (Active Comparator): Docetaxel 25 mg/m^2 IV over 30 minutes for 4 weeks with premedication with Dexamethasone, followed by 2 weeks off therapy.
  Interventions: Drug: Docetaxel; Drug: Dexamethasone
- Weekly Docetaxel + ZD1839 (Active Comparator): Docetaxel 25 mg/m^2 IV over 30 minutes for 4 weeks with premedication with Dexamethasone, followed by 2 weeks off therapy. ZD1839 250 mg by mouth daily, without break.
  Interventions: Drug: Docetaxel; Drug: ZD1839; Drug: Dexamethasone

INTERVENTIONS:
Drug: Docetaxel — 25 mg/m2 IV over 30 minutes for 4 weeks, followed by 2 weeks off therapy.
  Other Names: Taxotere
Drug: ZD1839 — 250 mg by mouth daily, without break.
  Other Names: Iressa; Gefitinib
  Arms: Weekly Docetaxel + ZD1839
Drug: Dexamethasone — Course #1: 3 doses of prophylactic Dexamethasone 4mg orally every 12 hours, starting the night before the Docetaxel infusion.
  Course #2: If no hypersensitivity reactions and no significant fluid retention during course 1, the Dexamethasone is reduced to 4mg orally twice daily on the day of therapy.
  Course #3 and subsequent courses: If no hypersensitivity reactions and no significant fluid retention during course 2, the Dexamethasone is reduced to 4mg orally one hour before treatment.

SUMMARY:
Primary Objective:

1. To compare the proportion of patients free from progression 9 months from the start of consolidation therapy with the combination of docetaxel and ZD1839 (Iressa) versus docetaxel alone. For the purposes of this protocol, "consolidation" therapy refers to treatment given at the time of maximal benefit from conventional front-line multi-agent chemotherapy.

Secondary Objective:

1. To compare time to progression (TTP), overall survival (OS) and cause-specific survival (CSS) in the two arms. For completeness, these will be reported both from the initiation of consolidation chemotherapy, and from the completion of induction chemotherapy.

DETAILED DESCRIPTION:
Docetaxel is a drug designed to help stop cancer cells from growing and dividing. ZD1839 is also a drug designed to block cancer cells from growing and dividing.

Before treatment starts, you will have a complete physical exam. Blood (2-3 tablespoons) and urine tests will be taken as part of the usual evaluation of liver, bone marrow, blood clotting ability, and kidney function. A chest x-ray and ECG (test to measure the electrical activity of the heart) will be done. You will have imaging studies such as a CT scan of the chest abdomen and pelvis and a bone scan to show the location of current tumors. If needed, an MRI scan of the brain will be done. This evaluation is considered standard. Women who are able to have children must have a negative blood pregnancy test. Patients who have a history of invasive tumors in their bladder, and who have not had a prior cystoscopy, must have a screening cystoscopy with an EUA (examination under anesthesia), to check the extent of disease in their bladder. An EUA of the bladder is a standard procedure for diagnosing and checking the status of bladder cancer.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive docetaxel alone. Participants in the other group will receive docetaxel plus ZD1839. There is an equal chance of being assigned to either group. Both you and the study doctor will know to which group you were assigned.

Docetaxel will be given through a catheter (a plastic tube) placed in a large vein in the chest or arm. The medication will be given over about thirty minutes one day each week for 4 weeks. This will be followed by a 2 week break. The 4 weeks of treatment and 2 weeks without treatment will be considered one course (6 weeks).

Dexamethasone will be given to decrease the risk of having an allergic reaction to the docetaxel. In the first cycle, you will receive 3 doses of dexamethasone by mouth every 12 hours starting the night before the docetaxel infusion. If you have no reaction, the dexamethasone will be decreased in Course 2 to one dose twice on the day of therapy. If there is no reaction in Course 2, the dexamethasone will be decreased further to 1 dose 1 hour before docetaxel treatment.

ZD1839 is a medication taken by mouth every day without break. Participants in the docetaxel plus ZD1839 group will take one ZD1839 tablet once a day at about the same time. You can take ZD1839 with or without food. If you forget to take a dose, take the last missed dose as soon as you remember, as long as it is at least 12 hours before the next dose is due. If it is less than 12 hours until the next dose, do not take the dose you have missed.

During treatment, you will have a weekly blood test (2-3 tablespoons) to measure bone marrow function. A physical exam and blood tests (2-3 tablespoons) will be repeated before each cycle of treatment. Imaging studies will be repeated at 9 months but may be performed sooner if you have symptoms that show your tumor may be getting worse. These scans are considered part of standard routine follow-up.

You will be on study as long as the tumor is not growing at a certain rate and there are no severe side effects. Therapy will be stopped and you may be taken off study early if one or both of these things occur. After 6 months, patients can choose to continue therapy if they wish. At the end of 4 cycles, you will have the option to continue your assigned therapy as long as it is tolerated and there is no evidence that the disease is getting worse. There is no maximum amount of time that you can receive treatment on this study.

After the study is complete, follow-up will be arranged at the discretion of your treating physician.

This is an investigational study. The FDA has authorized ZD1839 for research use only. A total of 90 patients may take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologic demonstration of metastatic or locally unresectable transitional cell carcinoma of the urothelium. Minor components (<50% overall) of variants such as glandular or squamous differentiation, or evolution to more aggressive phenotypes such as sarcomatoid of small cell change are acceptable. However, when these atypical histologies are dominant, other treatment approaches may be appropriate, and such patients are not eligible.
* All patients must have demonstrated some objective response to combination chemotherapy, and be clinically without progression since this response was appreciated. In general, patients will have been treated with at least two successive combination regimens in order to achieve maximum benefit from available chemotherapy.
* Patients who have not achieved a complete response to therapy must have received one of the chemotherapy regimens outlined in Appendix D prior to receiving consolidation therapy. Exceptions to this generalization would include patients with a near complete response to the first regimen given, or patients that are not fit for aggressive chemotherapy beyond an initially used regimen to which they responded. Patients must begin "consolidation" therapy within 6 weeks of the end of the last cycle of induction chemotherapy, and should begin as soon as possible.
* Zubrod performance status of 3 or better. If PS = 3 this must, in the opinion of the investigator, be secondary to the effects of induction chemotherapy and not the underlying cancer.
* Patients with a history of cardiac disease, or an ejection fraction (EF) less than 50% at the time of initiation of chemotherapy, must be demonstrated to have an ejection fraction of at least 40%. In addition, patients having received more than 250 mg/m^2 of doxorubicin during their induction phase, or who have EKG changes since initiation of chemotherapy must have an EF of at least 45%. Patients with no history of cardiac disease, a normal EKG and no more than 250 mg/m^2 of doxorubicin are not required to have an EF measurement.
* Provision of written informed consent.
* Women of childbearing potential must be willing to practice acceptable methods of birth control to prevent pregnancy.
* Males taking ZD1839 must also use birth control while taking the drug to avoid pregnancy in their partner.
* International normalized ratio (INR) elevations, bleeding, or both events have been reported in some patients taking warfarin. Patients taking warfarin with a target INR of > or = 2, should be monitored regularly (every week in the first cycle, with further monitoring based on the experience in the first cycle) for changes in prothrombin time (PT) or INR. Patients on prophylactic low dose warfarin (ie: 1-2 mg qd for central line thrombosis prophylaxis) do not require frequent monitoring.

Exclusion Criteria:

* Predominantly small cell histology.
* AST or conjugated bilirubin greater than twice the upper limit of normal.
* Serum creatinine greater than 2.5 mg/dL , or a creatinine clearance (either measured or estimated by Cockcroft formula) of less than 25 mL/min: creatinine clearance (CLcr) = [(140-age) x wt(kg)]/[72 xCreat (mg/dL)] (Multiply by 0.85 for females)
* Absolute neutrophil count (ANC) less than 1,000; Platelets less than 75,000.
* Prior (lifetime) cumulative exposure to doxorubicin greater than 400 mg/m^2.
* Pregnant and lactating women are excluded. Women of childbearing potential must have a negative pregnancy test prior to starting therapy.
* An active, or likely to become active, second malignancy.
* Known severe hypersensitivity to ZD1839 or any of the excipients of this product.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital of St. John's Wort
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment.
* Incomplete healing from previous oncologic or other major surgery
* Note that there is no requirement for measurable or evaluable disease. Evaluation of response to therapy is not an endpoint of this trial.
* Prior treatment with therapy which specifically targets the HER family of receptors.
* Patients with peripheral neuropathy > or = to grade 2 should be excluded. Patients may be included if their neuropathy has resolved to grade 1 by the time they are registered on the protocol.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease).
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: From April of 2004 to November of 2007, fifty patients with metastatic or surgically unresectable urothelial cancer were enrolled at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Weekly Docetaxel | Weekly Docetaxel + ZD1839
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Docetaxel | Weekly Docetaxel + ZD1839 | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 64 [51 to 76] | 62 [40 to 80] | 64 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 18 | 22
  Male | 21 | 7 | 28
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Progression 9 Months From Start of Consolidation Therapy
Description: The proportion of participants' progression free at 9 months compared between treatments using chi-square. Progressive disease was defined as at least a 25% increase from baseline, of the sum of the products of the two greatest dimensions of representative measurable lesions. Increasing severity in symptoms due to progressive tumor was also counted as progression even if they were not accompanied by an objective indicator on radiographic imaging. The development of any new measurable lesions was considered evidence of progressive cancer as well.
Time Frame: Assessment at 9 Months of therapy
Population: In order to test the trial hypotheses for the two cohorts progression at nine months, a sample size of 45 participants for each arm was required. Accrual was not met to assess the outcome hypotheses thus no participant analysis available.
Arm/Group | Weekly Docetaxel | Weekly Docetaxel + ZD1839
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Median Overall Survival
Description: Overall survival was summarized using the Kaplan-Meier estimation.
Time Frame: Baseline till participant death or end of follow-up period, assessed every 4 weeks, up to 5 years.
Population: Analysis by intent to treat population with all participants treated included.
Measure: Median (Full Range); unit: Months
Arm/Group | Weekly Docetaxel | Weekly Docetaxel + ZD1839
Number analyzed (Participants) | 25 | 25
Months | 18.0 [3.4 to 92] | 16.6 [3.9 to 95.9]

3. Secondary Outcome: Median Progression Free Survival From Trial Enrollment for Overall Study
Description: Progressive disease was defined as at least a 25% increase from baseline, of the sum of the products of the two greatest dimensions of representative measurable lesions. Increasing severity in symptoms due to progressive tumor was also counted as progression even if they were not accompanied by an objective indicator on radiographic imaging. The development of any new measurable lesions was considered evidence of progressive cancer as well.
Time Frame: From trial enrollment to disease progression or death, up to five years
Population: Analysis by intent to treat population with all participants treated included.
Measure: Median (Full Range); unit: Months
Arm/Group | Weekly Docetaxel | Weekly Docetaxel + ZD1839
Number analyzed (Participants) | 25 | 25
Months | 3.7 [0.7 to 10.4] | 4.4 [1.1 to 13.9]

ADVERSE EVENTS:
Time Frame: Clinical assessment at the end of each 6-week treatment where data on symptom status, pain medication use, and acute and cumulative toxicity recorded. Overall collection period: May 2004 to October 2013.
Arm/Group | Weekly Docetaxel | Weekly Docetaxel + ZD1839
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weekly Docetaxel (N=25) | Weekly Docetaxel + ZD1839 (N=25)
Rash (Skin and subcutaneous tissue disorders) | 0 | 6
Anemia (Blood and lymphatic system disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Dehydration (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysgeusia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Edema (Skin and subcutaneous tissue disorders) | 1 | 1
Fatigue (General disorders) | 6 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 1 | 2
Neuropathy (Nervous system disorders) | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Watery eyes (Eye disorders) | 0 | 2
Weakness (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes